CLINICAL TRIAL: NCT04933292
Title: A Randomised Clinical Trial Assessing the Efficacy and Safety of Mycophenolate Mofetil Versus Azathioprine for Induction of Remission in Treatment Primary Biliary Cholangitis-Autoimmune Hepatitis Overlap Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaoli Fan (Other)
Responsible Party: Sponsor-Investigator, Xiaoli Fan, Doctor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OS-2
Record Dates: First submitted 2020-05-01; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Autoimmune Hepatitis; Primary Biliary Cirrhosis
MeSH Terms: conditions — Hepatitis, Autoimmune; Liver Cirrhosis, Biliary | interventions — Methylprednisolone; Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone and Mycophenolate mofetil (Experimental)
  Interventions: Drug: Methylprednisolone and Mycophenolate mofetil
- Methylprednisolone and Azathioprine (Active Comparator)
  Interventions: Drug: Methylprednisolone and azathioprine

INTERVENTIONS:
Drug: Methylprednisolone and Mycophenolate mofetil — Methylprednisolone combination of mycophenolate mofetil
  Arms: Methylprednisolone and Mycophenolate mofetil
Drug: Methylprednisolone and azathioprine — Methylprednisolone combination of azathioprine
  Arms: Methylprednisolone and Azathioprine

SUMMARY:
Current standard therapy of primary biliary cholangitis-autoimmune hepatitis overlap syndrome(PBC-AIH overlap) consists of a combination of prednisolone and azathioprine. However, a significant proportion of patients may do not respond to, or is intolerant for azathioprine. Several studies have documented the efficacy and safety of mycophenolate mofetil(MMF) as second-line therapy for PBC-AIH overlap. However, robust evidence from a formal randomized clinical trial for the first-line immunosuppressor is in need.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years;
2. Diagnosed with PBC-AIH overlap syndrome according to Paris criteria;
3. Agreed to participate in the trial, and assigned informed consent;
4. The WBC count ≥2.5x10^9/L and platelet count ≥50x10^9/L.

Exclusion Criteria:

1. The presence of hepatitis A, B, C, D, or E virus infection;
2. Patients with presence of serious decompensated cirrhosis;
3. Patients have a history of glucocorticoid or immunosuppressant medication before enrollment;
4. Liver damage caused by other reasons: such as primary sclerosing cholangitis, non-alcoholic steatohepatitis, drug induced liver disease or Wilson disease.
5. Pregnant and breeding women;
6. Severe disorders of other vital organs, such as severe heart failure, cancer;
7. Parenteral administration of blood or blood products within 6 months before screening;
8. Recent treatment with drugs having known liver toxicity;
9. Taken part in other clinic trials within 6 months before enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Biochemical remission | 6 months
  The percentage of patients in remission, defined as normalization of serum transaminase and IgG levels after 6 months of treatment, per treatment group

SECONDARY OUTCOMES:
The level of IgG value in both groups | at 1 month
The level of IgG value in both groups | at 3-month
The level of IgG value in both groups | at 6-month
Adverse drug reactions | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan Univerisity, Chengdu, Sichuan, China